CLINICAL TRIAL: NCT06027515
Title: A Multimodal Prehabilitation Feasibility Study for Older Adult Patients at High Risk for Poor Postoperative Outcomes Prior to Esophageal Cancer Surgery
Brief Title: Esophageal Cancer Multimodal Prehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hassan Dashti, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-085
Record Dates: First submitted 2023-08-22; First posted 2023-09-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Cancer; Esophageal Neoplasms
Keywords: Esophageal Cancer; Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation Program (Experimental): 30 participants will be enrolled and will complete study procedures as follows:
  * Enrollment at least 4 weeks prior to esophageal cancer surgery.
  * In-person clinic visit with dietitian and physical therapist for assessments, and completion of baseline questionnaires with study coordinator.
  * Adherence to daily physical function, dietary, and sleep recommendations and consumption of 5-day immunonutrition supplement.
  * Regular electronic/phone-call check-ins with study staff.
  * Telehealth appointment with physical therapist and dietitian prior to surgery.
  * After surgery and during hospital admission, final visit with dietitian and physical therapist for assessments, and completion of questionnaires.
  * 6-month follow-up period.
  Interventions: Behavioral: Prehabilitation Program

INTERVENTIONS:
Behavioral: Prehabilitation Program — Multimodal prehabilitation program consisting of pre-surgical optimization of nutrition, physical function, and sleep health via individualized plans. Participants will also be supplied with Nestle Impact Advances Recovery Immunonutrition Drink.

SUMMARY:
The goal of this research study is to investigate the feasibility of implementing a prehabilitation program that aims to improve a patient's physical, nutritional, and sleep health before surgery in an older, at-risk group with esophageal cancer.

DETAILED DESCRIPTION:
This research study is to test whether a novel, 4-week surgical multimodal prehabilitation protocol is feasible in at-risk older adult patients who have previously undergone neoadjuvant chemotherapy or radiotherapy and are scheduled for surgical removal of esophageal cancer.

Research study procedures include screening for eligibility, clinic visits, questionnaires, blood tests, and Computed Tomography (CT) scans.

Participation in this research study is expected to last 7 months.

It is expected about 30 patients will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and over
* Adult male or non-pregnant female volunteers
* Completed neoadjuvant chemotherapy or radiotherapy for esophageal cancer
* At least four weeks to esophageal cancer surgery
* Without skin conditions that preclude wearing sensors
* Able to speak English and consent

Exclusion Criteria:

* Participants in any other interventional study that may bias results or limit study adherence during our study
* Dietary restrictions that prevent consumption of nutritional supplements
* Women who are pregnant, nursing, or at risk of becoming pregnant
* Profound physical disability (for example, quadriplegia) that precludes participation in any aerobic or strength training.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate (Feasibility) | At screening
  Number of eligible patients who enroll in study
Completion Rate (Feasibility) | 30 days
  Defined as the number of patients who complete study procedures.

SECONDARY OUTCOMES:
Nutrition Compliance Rate (Feasibility) | 5 days
  Comparison of number of nutritional supplements consumed compared to number of nutritional supplements prescribed as determined from daily check-ins. A cut-off value of 80% will be used to indicate compliance.
Physical Function Compliance Rate (Feasibility) | 30 days
  Comparison of the total minutes of physical function completed compared to the total minutes of physical function prescribed as determined from daily check-ins and wearable device. A cut-off value of 80% will be used to indicate compliance.
Sleep Health Compliance Rate (Feasibility) | 30 days
  Comparison of the average daily hours of sleep duration, minutes of wake after sleep onset, and variability in sleep timing, achieved compared to prescribed as determined from actigraphy. A cut-off value of 80% will be used to indicate compliance.
Actigraphy Compliance Rate (Feasibility) | 30 days
  Total daily hours of actiwatch/wearable device wear-time. A cut-off value of 80% will be used to indicate compliance.

OTHER OUTCOMES:
Sarcopenia | At baseline
  Assessed by baseline Computed Tomography (CT) scan of the thorax.
Malnutrition | At baseline visit and second measure at post-operative 1 day visit
  Assessed by the Perioperative Nutrition Screen (PONS) Risk Score, a modified version of the malnutrition universal screening tool, which determines the presence of nutrition risk based on BMI, recent body weight loss, decrement of dietary intake, and preoperative albumin concentration.
Patient-Reported Sleep Measures | At baseline visit and second measure at post-operative 1 day visit
  Assessed by the International Physical Activity Questionnaire (IPAQ), a 27-item self-reported measure of physical activity.
Hand Grip Test | At baseline visit and second measure at post-operative 1 day visit
  Assessed by change in baseline and post-operative Hand Grip tests using a hand-held dynamometer. An average score is calculated using measurements from both hands.
BMI | At baseline visit and second measure at post-operative 1 day visit
  Assessed by change in baseline and post-operative height and weight.
Energy expenditure | At baseline visit and second measure at post-operative 1 day visit
  Assessed by change in baseline and post-operative Metabolic Cart, or indirect calorimetry.
6-Minute Walk Test | At baseline visit and second measure at post-operative 1 day visit
  Assessed by a baseline and a post-operative 6-Minute Walk Test, a sub-maximal exercise test used to assess aerobic capacity and endurance.
Patient-Reported Measures on Physical Function Score | At baseline visit and second measure at post-operative 1 day visit
  Assessed by Activity Measure for Post-Acute Care (AM-PAC), a standardized assessment used to measure the physical function and functional status of patients. The AM-PAC consists of 13 tests that divided into lower and upper extremity function, gait and balance and activities of daily living and instrumental activities of daily living. Also assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF), a 45-item self-reported measure to evaluate physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Dashti, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation